CLINICAL TRIAL: NCT04096690
Title: The Efficacy and Safety of Anti-PD-1 Antibody in Combination With Pegaspargase in the Treatment of Newly Diagnosed, Stage III to IV Extranodal Natural Killer/T-Cell Lymphoma, Nasal Type
Brief Title: Anti-PD-1 Antibody Combined With Pegaspargase in the Treatment of Advanced Stage NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director，Hematology Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-NK-2019
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Nasal Type Extranodal NK/T-Cell Lymphoma
Keywords: Anti-PD-1 antibody; Nasal Type Extranodal NK/T-Cell Lymphoma; Complete response rate; Safety
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — pegaspargase; spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-PD-1 antibody plus pegaspargase (Experimental): Participants will receive induction treatment for six cycles of Anti-PD-1 antibody plus pegaspargase (21-day cycle) and Anti-PD-1 antibody monotherapy maintenance treatment for about 2 years (21-cycle)
  Interventions: Drug: Pegaspargase; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Pegaspargase — Pegaspargase 3750IU administered by intramuscular injection on Day 1 of each 21-day cycle for 6 cycles in induction treatment
Drug: Anti-PD-1 monoclonal antibody — Anti-PD-1 antibody 200mg administered intravenously (IV) on Day 2 of each 21-day cycle for 6 cycles in induction treatment Anti-PD-1 antibody 200mg administered intravenously (IV) on Day 1 of each 21-day cycle for up to 28 cycles in maintenance treatment
  Other Names: Tyvyt

SUMMARY:
This open-label, single arm study will evaluate the efficacy and safety of anti-PD-1 antibody in combination with pegaspargase in treatment of newly diagnosed advanced stage NK/T-cell lymphoma.

DETAILED DESCRIPTION:
Extranodal natural killer (NK)/T-cell lymphoma (ENKTL), nasal type, is a distinct and heterogeneous histopathologic subtype of non-Hodgkin lymphoma (NHL), accounting for 5%~10%. The frequency of ENKTL among NHL patients is significantly higher in Asia than in Western countries, with poor prognosis. L-asparaginase-based chemotherapy has improved the survival for these patients with advanced stage. However, there is no standard of care for those patients with advanced stage. Anti-PD-1 antibody has been proven its efficacy in relapsed or refractory NK/T cell lymphoma. This open-label, single arm study will evaluate the efficacy and safety of PD-1 antibody in combination with pegaspargase in treatment of newly diagnosed advanced stage NK/T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed NK/T cell lymphoma based on 2016 WHO classification
* Treatment naive
* Age > 18 years
* Advanced stage
* Must has measurable lesion in CT or PET-CT prior to treatment
* ECOG 0,1,2
* Informed consented

Exclusion Criteria:

* Aggressive NK/T-cell leukemia
* Has accepted PD-1,PD-L1 or PD-L2 antibody before
* Has accepted autologous Stem cell transplantation before
* History of malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix 3 years prior to study treatment
* Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
* Primary CNS lymphoma
* Lab at enrollment (Unless caused by lymphoma): Neutrophile<1.5*10^9/L ;Platelet<50*10^9/L; ALT or AST >3*ULN; Creatinine>2*ULN
* Other uncontrollable medical condition that may that may interfere the participation of the study
* Not able to comply to the protocol for mental or other unknown reasons Pregnant or lactation
* HIV infection
* HBV-DNA or HCV-RNA positive
* Diagnosed immunodeficiency or received systemic corticoid therapy 2 weeks prior to first dose.
* Received attenuated live vaccine 4 weeks prior to first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria and 2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy.

SECONDARY OUTCOMES:
Overall response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria and 2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy.
Progression free survival | Baseline up to data cut-off (up to approximately 4 years)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 4 years)
  Overall survival in the overall study population was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event.
Duration of response | Baseline up to data cut-off (up to approximately 4 years)
  Time from first occurrence of documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR. Tumor assessments were performed with PET-CT.
EBV-DNA load change | End of induction treatment (approximately 1 year)
  EBV-DNA load at each cycle for comparison
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Baseline up to data cut-off (up to approximately 4 years)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Core 30 (EORTC QLQ-C30) Domain Scores | Baseline (pre-dose [Hour 0] on Cycle1 Day1), Cycle3 Day 1, end of treatment (up to Month 6), every 3 months 1st year, every 6 months 2nd year, and 12 months thereafter up to data cut-off, up to approximately 4 years (cycle length = 21 days)
  The EORTC QLQ-C30 is a health-related quality of life questionnaire. A higher score indicates better quality of life, with changes of 5 to 10 points considered to be a minimally important difference to participants.
Treatment related mortality | Baseline up to data cut-off (up to approximately 4 years)
  Percentage of death related with treatment on the basis of investigator assessments

OTHER OUTCOMES:
Circulating free Deoxyribonucleic Acid (cfDNA) monitoring | Baseline up to data cut-off (up to approximately 4 years)
  CfDNA in peripheral blood assessed by local lab

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China